CLINICAL TRIAL: NCT01063166
Title: Collaboration on Alcohol Self Administration in Adolescents and Young Adults - Specific Aim 1: Assess the Initial Slope of Adolescent Drinking Trajectories, Beginning at the Age of Eighteen
Brief Title: Prospective Assessment of Adolescent Drinking Trajectories With Computer-Assisted Self-administration of Ethanol (CASE)
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Collaborators: Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: U01 AA017900 SA1; U01AA017900 (NIH)
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Alcoholism
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Computer-Assisted Self-administration of Ethanol (CASE)will be administered twice, at the ages 18 and 20, in a prospective study of 80 adolescents living in the Dresden area. The sample will be recruited for a differential family history of alcoholism (FHA) and gender, with inventories of alcohol use disorder (AUD) symptoms and personal recent drinking history (RDH) obtained prior to each CASE session.

ELIGIBILITY:
Inclusion Criteria:

* (a) male and female Caucasian volunteers aged 18 years/0 months to 19 years/11 months;
* (b) written informed consent by the subject;
* (c) habitual social drinking during the two months preceding participation, defined by at least one drinking day in any two weeks-interval;
* (d) at least one prior experience of alcohol intoxication
* (e) being able to abstain from tobacco use for four hours without developing nicotine withdrawal symptoms;
* (f) effective contraception in female participants;
* (g) consenting to abstain from any illegal substance use for 2 weeks prior to participation;
* (h) living within 15 km (9.5 miles) from downtown Dresden;
* (i) sufficient information concerning alcohol use in both parents and in at least four second-degree relatives

Exclusion Criteria:

* (a) prior medical treatment due to alcohol use;
* (b) current or prior history of any serious disease, including CNS, cardiovascular, respiratory, gastrointestinal, hepatic, renal, endocrine, alcohol or drug dependence, but not alcohol abuse;
* (c) current history of Axis-I psychiatric illness, including premenstrual dysphoric disorder;
* (d) current or prior history of alcohol-induced flushing reactions;
* (e) positive urine screen for cannabinoids, cocaine, amphetamines, opiates, or benzodiazepines;
* (f) light or non-drinkers: averaging less than 2 standard drinks per week in the preceding two months;
* (g) intention to become pregnant
* (h) pregnancy or positive urine pregnancy screening or breast-feeding;
* (i) any alcohol intake on the test day or the day before;
* (k) use of medications known to interact with alcohol within 2 weeks of the study;
* (l) positive hepatitis or HIV at screening, provided the subject consented to these tests

Ages: 18 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Residents living within 15 km (9.5 miles) from downtown Dresden
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2010-06; Primary Completion 2012-03 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Alcohol consumption | 2 years
  Alcohol consumption, as measured by a Timeline Followback Interview and experimental Self-Administration.

SECONDARY OUTCOMES:
Alcohol Use Disorders | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich S Zimmermann, Dr., Principal Investigator — Universitaetsklinikum Carl Gustav Carus at the Technische Universitaet Dresden
Locations (1):
- Universitaetsklinikum Carl Gustav Carus at the Technische Universitaet Dresden, Dresden, Saxony, Germany

REFERENCES:
- [Derived] Obst E, Bernhardt N, Gan G, Plawecki MH, O'Connor S, Smolka MN, Zimmermann US. Sensation seeking, impulsivity, and aggression moderate sex effects on adolescent laboratory binging. Psychol Addict Behav. 2021 Mar;35(2):208-214. doi: 10.1037/adb0000651. Epub 2020 Jun 25. PMID 32584051